CLINICAL TRIAL: NCT03820843
Title: Impact of Art Therapy on Brain Connectivity in Recent Post-Stroke Aphasia (ART-CONNECT)
Brief Title: Impact of Art Therapy on Brain Connectivity in Recent Post-Stroke Aphasia
Acronym: ART-CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP180312; N° IDRCB: 2018-A02462-53 (Other: ANSM)
Record Dates: First submitted 2019-01-10; First posted 2019-01-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Ischemic or Hemorrhagic Stroke
Keywords: brain connectivity; aphasia; art therapy; rehabilitation
MeSH Terms: conditions — Ischemia; Hemorrhagic Stroke; Aphasia | interventions — Art Therapy

STUDY DESIGN:
Intervention Model Description: The investigators will evaluate the reorganization of functional and structural brain connectivity maps before and after rehabilitation of aphasia with art therapy and standard orthophonic rehabilitation versus a control group that received only standard orthophonic rehabilitation.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single-blind: only the art therapist knows the randomization arm. The investigators involved in the outcomes assessement, will remain blinded with regard to the randomized treatment assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art therapy (Experimental): Art therapy and standard orthophonic rehabilitation
  Interventions: Other: Art therapy and standard orthophonic rehabilitation
- Control group (No Intervention): Only standard orthophonic rehabilitation

INTERVENTIONS:
Other: Art therapy and standard orthophonic rehabilitation — In addition to standard orthophonic rehabilitation, the patient will receive 12 sessions of art therapy
  Arms: Art therapy

SUMMARY:
A stroke located in the left parieto-temporal junction is associated, in aphasic right-handed patients, with a poor prognosis for language recovery. The role of the right hemisphere in recovering post-stroke aphasia is still controversial. Our hypothesis, based on recent work in imaging, is that early activation of the right hemisphere linked to the practice of the visual arts could facilitate language recovery in extended posterior left strokes that completely disrupt language areas.

DETAILED DESCRIPTION:
The investigators will evaluate, at inclusion and at 6 weeks, the reorganization of functional and structural brain connectivity maps before and after rehabilitation of aphasia with art therapy and standard orthophonic rehabilitation versus a control group that received only standard orthophonic rehabilitation.

The investigators will include all consecutive patients with recent ischemic or hemorrhagic stroke with unilateral lesion(s) of the parieto-temporal left junction present on the Diffusion MRI (DWI) performed in acute phase at 24-48h.

All patients will undergo 2 MRI with tensor diffusion sequences (structural connectivity) and fMRI (functional magnetic resonance imaging) resting state sequences (functional connectivity) at inclusion and 6 weeks after rehabilitation with or without art therapy.

The investigators aimed to demonstrate that early activation of the right hemisphere related to the practice of the visual arts could facilitate the recovery of language in later strokes completely disrupting the language areas of the left hemisphere.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recent ischemic or haemorrhagic stroke with unilateral lesion (s) of the parieto-temporal left junction present on the Diffusion MRI (DWI) performed in acute phase at 24-48h
* Post stroke delay of 15 days to 2 months
* Existence of moderate to severe phasic disorders on Aphasia Rapid Test score (ART, score> 6, scale of 26 items)
* Patient able to read and understand French
* Rightful
* Normal and corrected vision and hearing
* Absence of pre-existing degenerative neurological disorder
* Patient having signed his consent
* Age ≥ 18 years

Exclusion Criteria:

* Patients with contraindications to MRI or claustrophobic
* Patients under legal protection
* Patients with behavioral disorders or disabling neurovisual disorders making participation in art therapy impossible
* Mute patients, illiterate patients
* Patients leaving the neurological SSR department prematurely
* Patients not affiliated to a social security scheme
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
change from baseline measurement of white substance bundles volumes for structural connectivity at 6 weeks | from inclusion at 6 weeks
change from baseline measurement of synchrony amplitude of slow fluctuations for functional Connectivity at 6 weeks | from inclusion at 6 weeks

SECONDARY OUTCOMES:
change from baseline Aphasia at 6 weeks | from inclusion at 6 weeks
  The BDAE (Boston Diagnostic Aphasia Examination) score ranges from 0 to 5, with higher values indicating more severe impairment
change from baseline Aphasia at 6 weeks | from inclusion at 6 weeks
  The ART (Aphasia Rapid Test) score ranges from 0 to 26, with higher values indicating more severe impairment
change from baseline Anxiety and depression at 6 weeks | from inclusion and at 6 weeks
  The HADS (Hospital Anxiety and Depression Scale) scores ranges from 0 to 21 for both anxiety and depression scores, with higher values indicating more severe impairment
change from baseline Quality of life self-assessment at 6 weeks | from inclusion at 6 weeks
  Visual Analogic scale of patient quality of life is a 0% to 100% scale, with 100 indicating the best health status
Satisfaction self-assessment at 6 weeks | at 6 weeks only
  visual analogic scale of patient satisfaction is a 0 to 10 scale, with higher values indicating better satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Dupont, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Soins de Suite et Réadaptation, Paris, France

IPD SHARING:
Plan to Share IPD: No